CLINICAL TRIAL: NCT04446572
Title: Application of Lactobacillus Salivarius CECT5713 to Achieve Term Pregnancies in Women With Repetitive Abortion or Infertility of Unknown Origin by Microbiological and Immunological Modulation of the Vaginal Ecosystem
Brief Title: Application of Lactobacillus Salivarius CECT5713 in Infertility of Unknown Origin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Bisearch Life (Unknown); Centro de Diagnóstico Médico. Ayuntamiento de Madrid. (Unknown)
Responsible Party: Principal Investigator, Juan M. Rodríguez, Professor, Universidad Complutense de Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PREPROBIFERT01
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Abortion, Spontaneous; Abortion in First Trimester; Infertility Unexplained
Keywords: Infertility; Abortion
MeSH Terms: conditions — Abortion, Spontaneous; Infertility

STUDY DESIGN:
Intervention Model Description: Volunteers were classified into 3 groups. All women in the RA group (n = 21) had a history of recurrent miscarriage with three or more pregnancy losses during the first 12 weeks of pregnancy. All women of the INF group (n = 23) had a history of infertility (inability to conceive) despite being the recipients of assisted-reproduction techniques (ART) for at least three times, including two cycles, at least, of in vitro fertilization (IVF). Finally, the control group (n = 14) included fertile women having at least two children after uncomplicated term pregnancies. Starting at day 0, women of the RA and INF groups consumed (oral route) a daily sachet with ~50 mg of freeze-dried probiotic (~9 log10 CFU of L. salivarius CECT5713) for 6 months or until a diagnosis of pregnancy (whatever happened first).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Repetitive Abortion (RA) group (Experimental): Starting at day 0, women of the RA (n=21) group consumed (oral route) a daily sachet with ~50 mg of freeze-dried probiotic (~9 log10 CFU of L. salivarius CECT5713) for 6 months or until a diagnosis of pregnancy (whatever happened first).
  Interventions: Biological: Lactobacillus salivarius CECT5713
- Infertility (INF) group (Experimental): Starting at day 0, women of the INF group (n=23) consumed (oral route) a daily sachet with ~50 mg of freeze-dried probiotic (~9 log10 CFU of L. salivarius CECT5713) for 6 months or until a diagnosis of pregnancy (whatever happened first).
  Interventions: Biological: Lactobacillus salivarius CECT5713
- Control group (No Intervention): The control group (n = 14) included fertile women having at least two children after uncomplicated term pregnancies.

INTERVENTIONS:
Biological: Lactobacillus salivarius CECT5713 — Starting at day 0, women of the RA and INF groups consumed (oral route) a daily sachet with ~50 mg of freeze-dried probiotic (~9 log10 CFU of L. salivarius CECT5713) for 6 months or until a diagnosis of pregnancy (whatever happened first).
  Arms: Infertility (INF) group; Repetitive Abortion (RA) group

SUMMARY:
In this study, we aimed to assess the cervicovaginal environment (pH, Nugent score, soluble immune factors and bacterial profile) in women with reproductive failure because of either repetitive abortion or infertility of unknown origin and compare it to that of healthy fertile women. The second objective was to evaluate the ability of Lactobacillus salivarius CECT5713 to modulate such parameters and to increase pregnancy rates in women with reproductive failure. The administration of L. salivarius CECT5713 (~9 log10 colony-forming units (CFU)/day) for 6 months or until a diagnosis of pregnancy to women with reproductive failure resulted in an overall successful (term) pregnancy rate of 56%.

DETAILED DESCRIPTION:
In this study, we aimed to assess the cervicovaginal environment (pH, Nugent score, soluble immune factors and bacterial profile) in women with reproductive failure because of either repetitive abortion or infertility of unknown origin and compare it to that of healthy fertile women. The second objective was to evaluate the ability of Lactobacillus salivarius CECT5713 to modulate such parameters and to increase pregnancy rates in women with reproductive failure. Vaginal pH and Nugent score were higher in women with reproductive failure than in fertile women. Differences were also noted regarding soluble immune factors transforming growth factor beta (TGF-β) and vascular endothelial growth factor (VEGF). Their concentrations in cervicovaginal lavage samples were reduced by about one-half in women with reproductive failure compared to fertile women. Lactobacilli were detected in a higher proportion, and at a higher concentration and having different species profile, in fertile women than in women with repetitive abortion or infertility. The study of the vaginal microbiome revealed that samples from fertile women were characterized by the high abundance of Lactobacillus sequences, while in about one third of samples from women with reproductive failure DNA from this genus was practically absent while there was an abundance of that of Gardnerella and Bifidobacterium. Lactobacillus salivarius CECT5713 seemed to be a suitable candidate to modulate the cervicovaginal microbiota because of its acidifying capacity, adhesion to vaginal cells and co-aggregation with vaginal pathogens. The administration of L. salivarius CECT5713 (~9 log10 CFU/day) for 6 months or until a diagnosis of pregnancy to women with reproductive failure resulted in an overall successful (term) pregnancy rate of 56%. In addition, the probiotic intervention modified significantly key microbiological, biochemical and immunological parameters in women who got pregnant being their post-intervention values similar or close to those of fertile women. The high concentrations of L. salivarius and the detection of L. salivarius DNA in vaginal samples confirmed that the probiotic was able to reach the vaginal mucosa. In conclusion, L. salivarius CECT5713 has proved to be a good candidate to improve reproductive success in women with reproductive failure.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent miscarriage with three or more pregnancy losses during the first 12 weeks of pregnancy (RA group)
* Infertility (inability to conceive) despite being the recipients of ART for at least three times, including two cycles, at least, of in vitro fertilization (IVF) (INF group).
* Fertile women having at least two children after uncomplicated term pregnancies (Control group).

Exclusion Criteria:

* Antiphospholipid syndrome
* Hormonal therapy, antibiotics or probiotics in the 4 weeks previous to sampling.
* Lactose intolerance or cow's milk protein allergy (RA and INF groups)

Ages: 33 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The targets were abortion or female infertility of unknown origin
Enrollment: 58 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Pregnancies and successful pregnancies | 6 months
  Total number of pregnancies and number of pregnancies with delivery of a healthy baby

SECONDARY OUTCOMES:
Modification of the vaginal microbiota | 6 months
  Variation in the concentration of lactobacilli and other bacteria in cervicovaginal lavage samples
Vaginal immunomodulation | 6 months
  Variation in the concentration of TGF-β and VEGF in cervicovaginal lavage

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Rodríguez, PhD, Principal Investigator — Complutense University Madrid
Locations (1):
- Dpt. Nutricion, Bromatologia y Tecnologia de los Alimentos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Global and individual microbiological and immunological data will be available to other researchers once the study is published.
Supporting Information: Study Protocol, CSR
Time Frame: The data will be available to other researchers once the study is published.
Access Criteria: On request